CLINICAL TRIAL: NCT00712296
Title: Center for Chinese Herbal Therapy for Asthma. Project #2-Clinical Effect of a Chinese Herbal Therapy in Human Asthma-Phase II
Brief Title: Effectiveness of Chinese Herbal Therapy for Asthma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Xiu-Min Li, Professor, Pediatrics, Allergy and Immunology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 04-0206; P01AT002647-02 (NIH)
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Asthma
Keywords: Asthma; alternative medicine; complementary medicine; herbal therapy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ASHMI 4 (Experimental): ASHMI 4 capsules twice a day
  Interventions: Drug: ASHMI 4
- ASHMI 12 (Experimental): ASHMI 12 capsules twice a day
  Interventions: Drug: ASHMI 12
- Placebo (Placebo Comparator): Placebo 6 capsules twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASHMI 4 — 4 capsules orally twice a day
  Arms: ASHMI 4
Drug: ASHMI 12 — 12 capsules orally twice a day
  Arms: ASHMI 12
Drug: Placebo — Placebo 6 capsules twice a day
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of an anti-asthma herbal medicine intervention (ASHMI) in adult asthmatics

DETAILED DESCRIPTION:
Asthma is a major public health problem worldwide, particularly in westernized societies and has continued to increase in prevalence over the past two decades. Inhaled corticosteroids have become the first-line treatment for persistent asthma even though side effects have been reported. New asthma medications, including leukotriene inhibitors and anti-IgE, have shown limited benefits. Patients have increasingly turned to complementary and alternative medicine (CAM) for treatment of their asthma, despite the uncertainty of its benefits due a lack of well-controlled scientific studies.

We have developed a Chinese herbal formula composed of 3 herbs called ASHMI. It has been previously shown in murine studies that ASHMI (a formula containing Ling Zhi, Ku Shen and Gan Cao) has therapeutic effects on the major pathogenic mechanisms of asthma-airway hyperreactivity, pulmonary inflammation, and airway remodeling, as well as a down-regulating of TH2 response. A subsequent study in 91 asthmatic patients in Weifang, China found ASHMI to be a safe and effective alternative to prednisone for treating asthma and exhibited a beneficial effect on TH1 and TH2 balance. Additionally, a Phase I study conducted in the United States showed good tolerability to ASHMI. Based on these preliminary studies, we hypothesize that ASHMI will be a safe medication in patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ages 18 through 55 and otherwise in good health as determined by medical history and physical examination
* History of asthma documented by a physician for at least 6 months
* Females of childbearing potential must be sexually inactive or take effective birth control measures, as deemed appropriate by the investigator, for the duration of the study
* The subject agrees to participate in the study
* Subjects must have one of the following:
* one asthma-related unscheduled visit to an Emergency Department or clinic in the past 12 months
* One overnight hospitalization in the past 12 months
* Disturbed sleep more than twice in the past month
* Asthma symptoms ≥8 times in the past month
* use of a β2-agonist ≥8 times in the past month
* two short courses (3-7 days) of oral corticosteroids in the last 12 months
* FEV1 <80% predicted AND Use of inhaled corticosteroid (ICS) for at least 1 month prior to enrollment

Exclusion Criteria:

* Acute illness (such as cold, flu, etc.) within two weeks before the screening visit
* Any history of systemic disease that in the investigator's opinion would preclude the subject from participating in this study, including hepatitis virus infection
* History of chronic obstructive lung disease, emphysema, or other chronic respiratory condition
* Abnormal hepatic function (ALT/AST and bilirubin >1.25 x upper limit of normal)
* Abnormal bone marrow function (WBC <4 x 103/mm3; platelets <100 x 103/mm3; Hgb <11 g/dl)
* Abnormal renal function (BUN and creatinine >1.25 x upper limit of normal)
* Clinically significant abnormal electrocardiogram
* FEV1 <50% predicted
* Participation in another experimental therapy study within 30 days of this study
* History of alcohol or drug abuse
* Pregnant or lactating female subjects. Females of childbearing potential will need a negative serum pregnancy test at screening to be considered for this study
* Subjects receiving treatment with Omalizumab or immunotherapy for asthma

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2009-09-29 (Actual); Study Completion 2009-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Wisnivesky, MD, DrPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Wen MC, Wei CH, Hu ZQ, Srivastava K, Ko J, Xi ST, Mu DZ, Du JB, Li GH, Wallenstein S, Sampson H, Kattan M, Li XM. Efficacy and tolerability of anti-asthma herbal medicine intervention in adult patients with moderate-severe allergic asthma. J Allergy Clin Immunol. 2005 Sep;116(3):517-24. doi: 10.1016/j.jaci.2005.05.029. PMID 16159618

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 10/5/2006-3/12/2010
  Location: Mount Sinai School of Medicine, New York, NY
  Phase I Participants Screened 55 Consented 35 Excluded 13 Withdrawn 2
  Phase II Participants Screened 183 Consented 76 Excluded 19 Screen failed 11
Pre-assignment Details: Phase I: Time frame 1 week; Phase II: Time frame 28 weeks. Participants from Phase I were invited to participate in Phase II and were re-randomized to all three arms of Phase II.
Groups:
- Active, Phase I: Patients received 3 daily doses in which 2, 4 or 6 ASHMI capsules were administered twice a day for 7 days.
- Placebo, Phase I: Patients received placebo. (phase I)
- Active Phase II (ASHMI 4 Caps): Patients received active drug. 4 caps twice a day.
- Active, Phase II (ASHMI 12 Caps ): Patients received active drug. 12 caps twice a day.
- Placebo, Phase II: Patients received placebo. (phase II)
Period: Phase I ( 1 Week)
Arm/Group | Active, Phase I | Placebo, Phase I | Active Phase II (ASHMI 4 Caps) | Active, Phase II (ASHMI 12 Caps ) | Placebo, Phase II
Started | 12 | 8 | 0 | 0 | 0
Completed | 12 | 8 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Phase II (28 Weeks)
Arm/Group | Active, Phase I | Placebo, Phase I | Active Phase II (ASHMI 4 Caps) | Active, Phase II (ASHMI 12 Caps ) | Placebo, Phase II
Started | 0 | 0 | 15 | 16 | 15
Completed | 0 | 0 | 2 (ASHMI/Placebo was discontinued on 9/29/10.20 participants were re-randomized into the Phase II.) | 1 | 3
Not Completed | 0 | 0 | 13 | 15 | 12

BASELINE CHARACTERISTICS:
Population: ASHMI/Placebo was discontinued on 9/29/10. 20 participants were re-randomized into the Phase II.
Groups:
- Active, Phase I: Patients received 3 daily doses in which 2, 4, or 6 ASHMI capsules were administered twice a day for 7 days.
- Placebo, Phase I; Placebo, Phase II: Patients received placebo.
- Active, Phase II (ASHMI 4 Caps ): Patients received active drug, 4 caps twice a day
- Active, Phase II (ASHMI 12 Caps): Patients received active drug, 12 caps twice a day
- Total: Total of all reporting groups
Arm/Group | Active, Phase I | Placebo, Phase I | Active, Phase II (ASHMI 4 Caps ) | Active, Phase II (ASHMI 12 Caps) | Placebo, Phase II | Total
Number analyzed (Participants) | 12 | 8 | 15 | 16 | 15 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: ASHMI/Placebo was discontinued on 9/29/10.20 participants were re-randomized into the Phase II.
  years
    Phase 1: number analyzed (Participants) | 12 | 8 | 0 | 0 | 0 | 20
    Phase 1 | 32 (7) | 31 (9) |  |  |  | 31.6 (8.06)
    Phase 2: number analyzed (Participants) | 0 | 0 | 15 | 16 | 15 | 46
    Phase 2 |  |  | 44 (10) | 44 (8) | 40 (10) | 42.7 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants] — This includes the number of males and females for the randomized study population for Phase I and Phase II Population: ASHMI/Placebo was discontinued on 9/29/10.20 participants were re-randomized into the Phase II.
  Participants
    Phase 1: number analyzed (Participants) | 12 | 8 | 0 | 0 | 0 | 20
    Phase 1: Female | 9 | 5 |  |  |  | 14
    Phase 1: Male | 3 | 3 |  |  |  | 6
    Phase 2: number analyzed (Participants) | 0 | 0 | 15 | 16 | 15 | 46
    Phase 2: Female |  |  | 11 | 14 | 10 | 35
    Phase 2: Male |  |  | 4 | 2 | 5 | 11
Race/Ethnicity, Customized [Number; unit: participants] — Population: ASHMI/Placebo was discontinued on 9/29/10. 20 participants were re-randomized into the Phase II.
  participants
    Phase 1, White: number analyzed (Participants) | 12 | 8 | 0 | 0 | 0 | 20
    Phase 1, White | 3 | 6 |  |  |  | 23
    Phase 1, Black: number analyzed (Participants) | 12 | 8 | 0 | 0 | 0 | 20
    Phase 1, Black | 3 | 0 |  |  |  | 18
    Phase 1, Hispanic: number analyzed (Participants) | 12 | 8 | 0 | 0 | 0 | 20
    Phase 1, Hispanic | 5 | 2 |  |  |  | 19
    Phase 1, Asian: number analyzed (Participants) | 12 | 8 | 0 | 0 | 0 | 20
    Phase 1, Asian | 1 | 0 |  |  |  | 5
    Phase 1, Other: number analyzed (Participants) | 12 | 8 | 0 | 0 | 0 | 20
    Phase 1, Other | 0 | 0 |  |  |  | 1
    Phase 2, White: number analyzed (Participants) | 0 | 0 | 15 | 16 | 15 | 46
    Phase 2, White |  |  | 5 | 5 | 4 | 14
    Phase 2, Black: number analyzed (Participants) | 0 | 0 | 15 | 16 | 15 | 46
    Phase 2, Black |  |  | 6 | 7 | 2 | 15
    Phase 2, Hispanic: number analyzed (Participants) | 0 | 0 | 15 | 16 | 15 | 46
    Phase 2, Hispanic |  |  | 4 | 4 | 4 | 12
    Phase 2, Asian: number analyzed (Participants) | 0 | 0 | 15 | 16 | 15 | 46
    Phase 2, Asian |  |  | 0 | 0 | 4 | 4
    Phase 2, Other: number analyzed (Participants) | 0 | 0 | 15 | 16 | 15 | 46
    Phase 2, Other |  |  | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Glucose, Urea and Creatinine Phase I
Description: Summary of Laboratory data for Glucose(mg/dL), Urea(mg/dL) and Creatinine(mg/dL) in subjects enrolled in Phase 1
Time Frame: 1 week after receiving active drug or placebo
Population: For the Phase I study we used descriptive statistics to report the frequency of adverse events (AEs) among patients treated with ASHMI or placebo. Analysis was per intention to treat.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Active Phase I Baseline: Baseline results for patients on ASHMI.
- Active Phase I Post Treatment: Post Treatment results after 1 week for patients on ASHMI.
- Placebo Phase I Baseline: Baseline results for participants who received placebo.
- Placebo Phase I Post Treatment: Post Treatment results for participants who received placebo.
Arm/Group | Active Phase I Baseline | Active Phase I Post Treatment | Placebo Phase I Baseline | Placebo Phase I Post Treatment
Number analyzed (Participants) | 12 | 12 | 8 | 8
mg/dL
  Glucose | 81 (12) | 79 (9) | 75 (14) | 71 (7)
  Urea | 13 (3) | 13 (3) | 16 (4) | 17 (5)
  Creatinine | 0.8 (0.2) | 0.8 (0.2) | 0.9 (0.1) | 0.9 (0.2)

2. Primary Outcome: Sodium, Potassium, Chloride and CO2 Phase I
Description: Summary of Laboratory data for Sodium(meq/L), Potassium(meq/L), Chloride(meq/L) and CO2 (meq/L) in subjects enrolled in Phase 1
Time Frame: 1 week after receiving active drug or placebo
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meq/L
Arm/Group | Active Phase I Baseline | Active Phase I Post Treatment | Placebo Phase I Baseline | Placebo Phase I Post Treatment
Number analyzed (Participants) | 12 | 12 | 8 | 8
meq/L
  Sodium (meq/L) | 139 (2) | 140 (2) | 139 (3) | 139 (1)
  Potassium (meq/L) | 4 (0.3) | 4 (0.4) | 4 (0.4) | 4 (0.2)
  Chloride (meq/L) | 103 (2) | 103 (1) | 102 (1) | 102 (2)
  Carbon dioxide (meq/L) | 24 (3) | 23 (2) | 24 (2) | 24 (2)

3. Primary Outcome: Serum Glutamic Pyruvic Transaminase and Serum Glutamic Oxaloacetic Transaminase in Phase I
Description: Summary of Laboratory data for Serum glutamic pyruvic transaminase and Serum glutamic oxaloacetic transaminase in subjects enrolled in Phase 1
Time Frame: 1 week after receiving active drug and placebo
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Active Phase I Baseline | Active Phase I Post Treatment | Placebo Phase I Baseline | Placebo Phase I Post Treatment
Number analyzed (Participants) | 12 | 12 | 8 | 8
IU/L
  Serum glutamic pyruvic transaminase (SGPT) | 19 (8) | 20 (8) | 21 (9) | 20 (9)
  Serum glutamic oxaloacetic transaminase (SGOT) | 20 (4) | 20 (7) | 24 (8) | 24 (10)

4. Primary Outcome: Laboratory Results for White Blood Cell, Hemoglobin and Platelet in Phase I
Description: Summary of Laboratory data for White Blood Cell(cells*10^3/uL), Hemoglobin(cells*10^3/uL) and Platelet(cells*10^3/uL)in subjects enrolled in Phase 1
Time Frame: 1 week after receiving active drug and placebo
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells*10^3/uL
Arm/Group | Active Phase I Baseline | Active Phase I Post Treatment | Placebo Phase I Baseline | Placebo Phase I Post Treatment
Number analyzed (Participants) | 12 | 12 | 8 | 8
cells*10^3/uL
  White Blood Cell | 7 (2) | 7 (1) | 7 (2) | 7 (1)
  Platelet | 292 (81) | 238 (123) | 281 (60) | 273 (64)

5. Primary Outcome: Hemoglobin Laboratory Results in Phase I
Description: Summary of hemoglobin as Outcome measures included laboratory data for subjects enrolled in Phase 1
Time Frame: 1 week
Population: For the Phase I study descriptive statistics were used to report the frequency of adverse events (AEs) among patients treated with ASHMI or placebo. Analysis was per intention to treat.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Active Phase I Baseline | Active Phase I Post Treatment | Placebo Phase I Baseline | Placebo Phase I Post Treatment
Number analyzed (Participants) | 12 | 12 | 8 | 8
g/dL | 13 (0.9) | 13 (1) | 14 (2) | 14 (1)

6. Primary Outcome: Laboratory Results for Glucose, Urea, Creatinine, Bilirubin Total and Bilirubin Direct Phase II Study
Description: Summary of Laboratory data for Glucose(mg/dL), Urea(mg/dL), Creatinine(mg/dL), Bilirubin Total(mg/dL) and Bilirubin Direct(mg/dL)in subjects in Phase II
  Limited to Measurements before discontinuation of ASHMI treatment
Time Frame: 28 weeks
Population: The Phase II study was terminated in September 2009 before the planned enrollment of 50 subjects was completed. As of September 29, 2009, the trial was discontinued in accordance with recommendations of the Data Safety Monitoring Board (DSMB).
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Placebo Phase II Baseline: Patients received placebo. at baseline.
- Active Phase II (ASHMI 4 Caps) Baseline: Patients received active drug. 4 caps twice a day. at baseline.
- Active Phase II (ASHMI 12 Caps) Baseline: Patients received active drug. 12 caps twice a day. at baseline.
- Placebo Phase II Visit 5: Patients received placebo. at visit 5.
- Active Phase II (ASHMI 4 Caps) Visit 5: Patients received active drug. 4 caps twice a day. at visit 5.
- Active Phase II (ASHMI 12 Caps) Visit 5: Patients received active drug. 12 caps twice a day. at visit 5.
- Placebo Phase II Visit 10: Patients received placebo. at visit 10.
- Active Phase II (ASHMI 4 Caps) Visit 10: Patients received active drug. 4 caps twice a day. at visit 10.
- Active Phase II (ASHMI 12 Caps) Visit 10: Patients received active drug. 12 caps twice a day. at visit 10.
Arm/Group | Placebo Phase II Baseline | Active Phase II (ASHMI 4 Caps) Baseline | Active Phase II (ASHMI 12 Caps) Baseline | Placebo Phase II Visit 5 | Active Phase II (ASHMI 4 Caps) Visit 5 | Active Phase II (ASHMI 12 Caps) Visit 5 | Placebo Phase II Visit 10 | Active Phase II (ASHMI 4 Caps) Visit 10 | Active Phase II (ASHMI 12 Caps) Visit 10
Number analyzed (Participants) | 15 | 15 | 16 | 10 | 11 | 10 | 3 | 2 | 1
mg/dL
  Glucose | 85 (28.4) | 79.1 (12.1) | 77.1 (12.8) | 99.9 (45.9) | 77.6 (8.8) | 72.5 (12.6) | 92.0 (12.0) | 95.0 (38.2) | 101.0
  Urea | 14.8 (4.1) | 13.3 (5.4) | 14.1 (5.4) | 13.9 (2.6) | 13.3 (2.5) | 14.2 (4.2) | 15.0 (2.6) | 15.0 (8.5) | 18.0
  Creatinine | 0.9 (0.2) | 0.8 (0.2) | 0.8 (0.1) | 0.8 (0.1) | 0.9 (0.3) | 0.9 (0.2) | 1.0 (0.1) | 0.9 (0.1) | 0.3
  Bilirubin Total | 0.4 (0.2) | 0.4 (0.2) | 0.4 (0.2) | 0.5 (0.2) | 0.4 (0.2) | 0.3 (0.1) | 0.4 (0.2) | 0.4 (0.2) | 0.2
  Bilirubin Direct | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.1) | 0.1 (0.0) | 0.1

7. Primary Outcome: Laboratory Results for Sodium,Potassium, Chloride and Bicarbonate in Phase II Study
Description: Summary of Laboratory data for Sodium(meq/L), Potassium(meq/L), Chloride(meq/L) and Bicarbonate(meq/L)in subjects in Phase II
  Limited to Measurements before discontinuation of ASHMI treatment
Time Frame: 28 weeks
Population: The Phase II study was terminated in September 2009 before the planned enrollment of 50 subjects was completed.
Measure: Mean (Standard Deviation); unit: meq/L
Groups:
- Placebo Phase II Baseline: Patients received placebo at baseline
- Active Phase II (ASHMI 4 Caps ) Baseline: Patients received active drug. 4 caps twice a day at baseline
- Active Phase II (ASHMI 12 Caps) Baseline: Patients received active drug. 12 caps twice a day. Baseline
- Active Phase II (ASHMI 12 Caps) Visit 10: Patients received active drug. 12 caps a day. at visit 10.
Arm/Group | Placebo Phase II Baseline | Active Phase II (ASHMI 4 Caps ) Baseline | Active Phase II (ASHMI 12 Caps) Baseline | Placebo Phase II Visit 5 | Active Phase II (ASHMI 4 Caps) Visit 5 | Active Phase II (ASHMI 12 Caps) Visit 5 | Placebo Phase II Visit 10 | Active Phase II (ASHMI 4 Caps) Visit 10 | Active Phase II (ASHMI 12 Caps) Visit 10
Number analyzed (Participants) | 15 | 15 | 16 | 10 | 11 | 10 | 3 | 2 | 1
meq/L
  Sodium | 140.6 (1.6) | 140.3 (1.9) | 140.5 (2.3) | 139.5 (2.1) | 140.1 (2.2) | 139.6 (2.5) | 139.7 (1.5) | 140 (1.4) | 140.0
  Potassium | 3.9 (0.4) | 4.1 (0.2) | 4.1 (0.3) | 4.1 (0.3) | 4.1 (0.1) | 4.1 (0.3) | 4.2 (0.6) | 4.1 (0.5) | 3.8
  Chloride | 102.5 (2.2) | 102.6 (1.9) | 102.6 (2.5) | 102.4 (2.2) | 102.9 (3.2) | 102.3 (3.5) | 102.3 (0.6) | 101.5 (2.1) | 108.0
  Bicarbonate | 27.2 (2.7) | 26.7 (2.5) | 27.5 (1.6) | 25.8 (2.4) | 26.2 (2.0) | 26.2 (1.7) | 27.1 (1.6) | 26.3 (2.9) | 19.2

8. Primary Outcome: Laboratory Results for Alkaline Phosphatase,Serum Glutamic Pyruvic Transaminase and Serum Glutamic Oxaloacetic Transaminase in Phase II Study
Description: Summary of Laboratory data for Alkaline phosphatase(IU/L),Serum glutamic pyruvic transaminase(IU/L)and Serum glutamic oxaloacetic transaminase(IU/L) in subjects in Phase II study
  Limited to Measurements before discontinuation of ASHMI treatment
Time Frame: 28 weeks
Population: The Phase II study was terminated in September 2009 before the planned enrollment of 50 subjects was completed. As of September 28, 2009, the trial was discontinued in accordance with recommendations of the Data Safety Monitoring Board (DSMB).
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Placebo Phase II Baseline | Active Phase II (ASHMI 4 Caps) Baseline | Active Phase II (ASHMI 12 Caps) Baseline | Placebo Phase II Visit 5 | Active Phase II (ASHMI 4 Caps) Visit 5 | Active Phase II (ASHMI 12 Caps) Visit 5 | Placebo Phase II Visit 10 | Active Phase II (ASHMI 4 Caps) Visit 10 | Active Phase II (ASHMI 12 Caps) Visit 10
Number analyzed (Participants) | 15 | 15 | 16 | 10 | 11 | 10 | 3 | 2 | 1
IU/L
  Alkaline phosphatase | 76.0 (22.2) | 91.3 (23.0) | 76.6 (24.7) | 81.1 (24.8) | 29.7 (25.7) | 83.2 (25.0) | 61.7 (18.5) | 98.0 (5.7) | 78.0
  Serum glutamic pyruvic transaminase (SGPT) | 23.9 (11.6) | 21.9 (18.2) | 21.3 (9.4) | 26.9 (11.9) | 22.0 (11.0) | 22.5 (8.6) | 24.3 (7.4) | 14.5 (4.9) | 32.0
  Serum glutamic oxaloacetic transaminase (SGOT) | 24.5 (8.4) | 22.0 (9.3) | 24.7 (7.3) | 24.8 (8.1) | 25.8 (9.6) | 25.6 (8.7) | 25.3 (8.9) | 21.0 (7.1) | 30.0

9. Primary Outcome: Laboratory Results for White Blood Cell Count and Platelet in Subjects in Phase II Study
Description: Summary of Laboratory data for White Blood Cell Count(cells*10^3/uL) and Platelet (cells*10^3/uL)in Phase II study
  Limited to Measurements before discontinuation of ASHMI treatment
Time Frame: 28 weeks
Population: The Phase II study was terminated in September 2009 before the planned enrollment of 50 subjects was completed. As of September 28, 2009,the trial was discontinued in accordance with recommendations of the Data Safety Monitoring Board (DSMB).
Measure: Mean (Standard Deviation); unit: cells*10^3/uL
Arm/Group | Placebo Phase II Baseline | Active Phase II (ASHMI 4 Caps) Baseline | Active Phase II (ASHMI 12 Caps) Baseline | Placebo Phase II Visit 5 | Active Phase II (ASHMI 4 Caps) Visit 5 | Active Phase II (ASHMI 12 Caps) Visit 5 | Placebo Phase II Visit 10 | Active Phase II (ASHMI 4 Caps) Visit 10 | Active Phase II (ASHMI 12 Caps) Visit 10
Number analyzed (Participants) | 15 | 15 | 16 | 10 | 11 | 10 | 3 | 2 | 1
cells*10^3/uL
  White Blood Cell Count | 7.2 (2.3) | 7.6 (2.6) | 7.2 (1.4) | 6.5 (2.1) | 7.5 (2.7) | 6.8 (1.9) | 7.9 (2.7) | 9.4 (0.7) | 6.2
  Platelet | 254.5 (74.6) | 268.2 (49.0) | 267.1 (89.5) | 275.0 (86.3) | 283.3 (58.5) | 275.6 (119.6) | 280.0 (133.8) | 348.5 (29.0) | 269.0

10. Primary Outcome: Laboratory Results for Hemoglobin in Subjects in Phase II Study
Description: Summary of Laboratory data for hemoglobin(g/dL)in subjects in Phase II study.
  Limited to Measurements before discontinuation of ASHMI treatment
Time Frame: 28 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Active Phase II (ASHMI 12 Caps) Baseline: Patients received active drug.12 caps twice a day. at baseline.
- Placebo Phase II Visit 10: Patients received placebo. at day 10.
- Active Phase II (ASHMI 12 Caps) Visit 10: Patients received active drug.12 caps twice a day. at visit 10.
Arm/Group | Placebo Phase II Baseline | Active Phase II (ASHMI 4 Caps) Baseline | Active Phase II (ASHMI 12 Caps) Baseline | Placebo Phase II Visit 5 | Active Phase II (ASHMI 4 Caps) Visit 5 | Active Phase II (ASHMI 12 Caps) Visit 5 | Placebo Phase II Visit 10 | Active Phase II (ASHMI 4 Caps) Visit 10 | Active Phase II (ASHMI 12 Caps) Visit 10
Number analyzed (Participants) | 15 | 15 | 16 | 10 | 11 | 10 | 3 | 2 | 1
g/dL | 13.5 (1.4) | 13.5 (1.6) | 12.8 (1.2) | 13.9 (1.2) | 13.7 (1.4) | 12.9 (1.5) | 13.7 (1.7) | 13.9 (1.5) | 14.3

ADVERSE EVENTS:
Time Frame: Phase I: 1 week Phase II: 28 weeks
Groups:
- Active Phase I (ASHMI 2 Caps Twice a Day): Patients received 2, 4, or 6 ASHMI capsules were administered twice daily for 7 days.
- Placebo Phase I (2 Caps Twice a Day): Patients received placebo. 2 caps twice a day.
- Active Phase I (ASHMI 4 Caps): Patients received active drug. 4 caps twice a day.
- Placebo Phase I (4 Caps Twice a Day): Patients received placebo. 4 caps twice a day.
- Active Phase I (ASHMI 6 Caps): Patients received active drug. 6 caps twice a day.
- Placebo Phase I; Placebo Phase II: Patients received placebo.
- Active Phase II (ASHMI 4 Caps Twice a Day): Patients received active drug.Based on revised adverse event criteria on January 2010.
- Active Phase II (ASHMI 12 Caps): Patients received active drug. 12 caps twice a day.
Arm/Group | Active Phase I (ASHMI 2 Caps Twice a Day) | Placebo Phase I (2 Caps Twice a Day) | Active Phase I (ASHMI 4 Caps) | Placebo Phase I (4 Caps Twice a Day) | Active Phase I (ASHMI 6 Caps) | Placebo Phase I | Active Phase II (ASHMI 4 Caps Twice a Day) | Active Phase II (ASHMI 12 Caps) | Placebo Phase II
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 0/4 | 0/4 | 0/4 | 0/2 | 0/15 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 2/4 | 2/2 | 1/4 | 2/4 | 1/4 | 1/2 | 2/15 | 2/16 | 3/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Phase I (ASHMI 2 Caps Twice a Day) (N=4) | Placebo Phase I (2 Caps Twice a Day) (N=2) | Active Phase I (ASHMI 4 Caps) (N=4) | Placebo Phase I (4 Caps Twice a Day) (N=4) | Active Phase I (ASHMI 6 Caps) (N=4) | Placebo Phase I (N=2) | Active Phase II (ASHMI 4 Caps Twice a Day) (N=15) | Active Phase II (ASHMI 12 Caps) (N=16) | Placebo Phase II (N=15)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body aches and fatigue associated with subject's typical prementrual syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient upper extremity itchiness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Insomnia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased total serum bicarbonate level (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back muscle injury (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glucosuria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased Glucose Level (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Decreased Hemoglobin Level (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Decreased White Blood Cell Count (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Emergency room visit for asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Unscheduled physician visit for asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Electrocardiogram changes (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Trichomonas in urine (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased Alkaline Phosphatase (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Increased Creatine (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal symptoms (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated Liver Enzymes (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The Phase II study was stopped after 46 subjects were randomized. Since the number of subjects and the follow-up information did not provide adequate power, all statistical analysis plan was changed to descriptive summaries for each group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No